CLINICAL TRIAL: NCT02655419
Title: A PHASE IIA PROSPECTIVE, OPEN-LABEL, MULTICENTER STUDY TO DETERMINE THE PHARMACOKINETICS (PK) AND SAFETY AND TOLERABILITY OF AZTREONAM-AVIBACTAM (ATM-AVI) FOR THE TREATMENT OF COMPLICATED INTRA-ABDOMINAL INFECTIONS (CIAIS) IN HOSPITALIZED ADULTS
Brief Title: Determine the PK and Safety and Tolerability of ATM-AVI for the Treatment of cIAIs in Hospitalized Adults (REJUVENATE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4910C00009; C3601001 (Other: Alias Study Number); 2015-002726-39 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2016-01-14 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Complicated Intra-Abdominal Infections, cIAIs
Keywords: cIAIs in hospitalized adults
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATM-AVI + Metronidazole (Experimental): Aztreonam-avibactam + metronidazole
  Interventions: Drug: ATM-AVI; Drug: Metronidazole

INTERVENTIONS:
Drug: ATM-AVI — Cohort 1:
  (Creatinine clearance > 50 mL/min)6500mg ATM/1777mg AVI on day 1 followed by total daily dose of 6000mg ATM/1640mg AVI
  Cohorts 2 and 3:
  (Creatinine clearance > 50 mL/min) As above, or: 6500 mg ATM/2167 mg on Day 1 followed by a total daily dose of 6000 mg ATM/2000 m AVI
  (Creatinine clearance 31 - 50 mL/min) 4250 mg ATM/1162 mg AVI on Day 1 followed by total daily dose 3000 mg ATM/820 mg AVI, or:
  4250 mg ATM/1417 mg AVI on Day 1 followed by total daily dose 3000 mg ATM/1000 mg AVI
Drug: Metronidazole — Metronidazole 500mg infused over 1 hour every 8 hours

SUMMARY:
Determine the PK and safety and tolerability of aztreonam-avibactam (ATM-AVI) in the treatment of hospitalized adults with cIAI

DETAILED DESCRIPTION:
A Phase IIa prospective, open-label, multicenter study to determine the pharmacokinetics (PK) and safety and tolerability of aztreonam-avibactam (ATM-AVI) for the treatment of complicated Intra-Abdominal Infections (cIAIs) in hospitalized adults.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Male or female from 18 to 90 years
3. Female patients are authorized to participate in this clinical study if criteria concerning pregnancy avoidance stated in the protocol are met
4. Diagnosis of cIAI

   EITHER:

   Intra-operative/postoperative enrolment with visual confirmation of cIAI. OR Preoperative enrollment with evidence of systemic inflammatory response, physical and radiological findings consistent with cIAI; confirmation of cIAI at time of surgery within 24 hours of study entry
5. Patients who failed prior antibacterial treatment for their current cIAI can be enrolled but must:

   * Have a known or suspected pathogen causing cIAI that is resistant to the prior therapy
   * Require surgical intervention.
6. Patient must have or will have a surgical intervention within 24 hours (before or after) the administration of the first dose of study drug

Exclusion criteria:

1. Involvement in the planning and/or conduct of the study
2. Patient has been previously enrolled in this study, previously treated with ATM-AVI or previously participated in an investigational study containing AVI
3. Patient has participated or intends to participate in any other clinical study that involves the administration of a study drug during the course of the study, or during the 30 days prior to study start.
4. History of serious allergy, hypersensitivity (eg, anaphylaxis), or any serious reaction to aztreonam, carbapenem,monobactam or other β-lactam antibiotics, avibactam, nitroimidazoles or metronidazole, or any of the excipients of the study drugs
5. Diagnosis of abdominal wall abscess; small bowel obstruction or ischemic bowel disease without perforation; traumatic bowel perforation with surgery within 12 hours of diagnosis; perforation of gastroduodenal ulcer with surgery within 24 hours of diagnosis primary etiology is not likely to be infectious
6. Simple cholecystitis, gangrenous cholecystitis without rupture, simple appendicitis, acute suppurative cholangitis, infected necrotizing pancreatitis, pancreatic abscess or ischaemic/necrotic intestine without perforation
7. Staged abdominal repair (STAR), open abdomen technique or where infection source control is not likely to be achieved; unlikely to solely respond to antimicrobial therapy
8. Infection due to a pathogen that is unlikely to respond to ATM-AVI plus metronidazole
9. Rapidly progressive or terminal illness
10. Systemic antibacterial agents received within the 72- hour period prior to study entry, unless:

    1. A new infection and no more than 24 hours of prior antibiotic treatment received within the 72 hour period prior to study entry or
    2. Patient is considered to have failed the previous treatment
11. Concurrent infection that may interfere with the evaluation of clinical cure for the study therapy
12. requirement for effective concomitant systemic antibacterials or antifungals
13. Creatinine clearance ≤30 ml/min or requirement for renal replacement therapy
14. Acute hepatitis in the prior 6 months, chronic hepatitis, cirrhosis, acute hepatic failure, or acute decompensation of chronic hepatic failure
15. Hepatic disease as indicated by AST or ALT >3 × ULN. Patients with AST and/or ALT >3 × ULN and < 5 × ULN are eligible if acute, not accompanied by a total bilirubin ≥ 2xULN and documented by the investigator as being directly related to cIAI.
16. Patient has a total bilirubin >3 × ULN, unless isolated hyperbilirubinemia is directly related to cIAI or due to known Gilbert's disease
17. ALP >3 × ULN. Patients with values >3 × ULN and <5 x ULN are eligible if acute and directly related to the infectious process being treated.
18. Immunocompromising illness
19. Active Clostridium difficile associated diarrhoea
20. Any other condition that may confound the results of the study or pose additional risks
21. Do not resuscitate order
22. Absolute neutrophil count <1000/μL
23. Hematocrit <25% or hemoglobin <8 gm/dL.
24. Platelet count <75,000/μL.
25. Currently receiving probenecid.
26. Pregnant or breastfeeding or if of child bearing potential, not using a medically accepted effective method of birth control.
27. Unlikely to comply with protocol,
28. Currently receiving anti-convulsant therapy to prevent recurrence of a past history of seizures.
29. Prior liver, pancreas or small-bowel transplant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Oliver Cornely, Principal Investigator — Clinical Trials Centre Cologne
Locations (11):
- France (2):
  - University Hospital C., Lille
  - CHU Limoges, Limoges
- Germany (2):
  - Universitaetsklinikum Koeln Innere Medizin I, Cologne
  - Universitaetsklinikum Schleswig-Holstein, Klinik fuer Infektiologie und Mikrobiologie, DZIF-CTU, Lübeck
- Spain (7):
  - Hospital Universitario Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Son Espases, Palma de Mallorca, ISLA Baleares
  - Hospital Universitari del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Mutua de Tarrasa, Terrassa

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Das S, Riccobene T, Carrothers TJ, Wright JG, MacPherson M, Cristinacce A, McFadyen L, Xie R, Luckey A, Raber S. Dose selection for aztreonam-avibactam, including adjustments for renal impairment, for Phase IIa and Phase III evaluation. Eur J Clin Pharmacol. 2024 Apr;80(4):529-543. doi: 10.1007/s00228-023-03609-x. Epub 2024 Jan 22. PMID 38252170
- [Derived] Jimenez-Rodriguez RM, Martin-Gutierrez G, Jimenez-Jorge S, Rosso-Fernandez CM, Tallon-Aguilar L, Roca-Oporto C, Padillo J, Luckey A, Cano A, Lopez-Ruiz J, Gomez-Zorrilla S, Bonnin-Pascual J, Boix-Palop L, Montejo JM, Torre-Cisneros J, Cisneros JM. Factors associated with recruitment success in the phase 2a study of aztreonam-avibactam development programme: a descriptive qualitative analysis among sites in Spain. BMJ Open. 2022 Feb 3;12(2):e051187. doi: 10.1136/bmjopen-2021-051187. PMID 35115349
- [Derived] Cornely OA, Cisneros JM, Torre-Cisneros J, Rodriguez-Hernandez MJ, Tallon-Aguilar L, Calbo E, Horcajada JP, Queckenberg C, Zettelmeyer U, Arenz D, Rosso-Fernandez CM, Jimenez-Jorge S, Turner G, Raber S, O'Brien S, Luckey A; COMBACTE-CARE consortium/REJUVENATE Study Group. Pharmacokinetics and safety of aztreonam/avibactam for the treatment of complicated intra-abdominal infections in hospitalized adults: results from the REJUVENATE study. J Antimicrob Chemother. 2020 Mar 1;75(3):618-627. doi: 10.1093/jac/dkz497. PMID 31828337
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=D4910C00009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at 11 centers in 3 countries from 19-May-2016 to 26-Oct-2017.
Groups:
- Aztreonam-Avibactam(ATM-AVI)+Metronidazole:Low AVI Dose Cohort: Participants with normal renal function or mild renal impairment (Creatinine clearance [CrCl] greater than[>] 50 milliliter per minute [mL/min]), received intravenous (IV) infusion of 500 milligram (mg) ATM plus 137 mg AVI over 30 minutes as loading dose, followed by maintenance infusions of 1500 mg ATM plus 410 mg AVI, over a 3 hour period every 6 hours, for a minimum of 5 days and up to maximum of 14 days. Participants also received 1 hour IV infusion of 500 mg metronidazole, every 8 hrs after first ATM-AVI maintenance infusion for a minimum of 5 days and up to maximum of 14 days. All study therapies could be discontinued (after at least 5 full days of IV therapy) at the discretion of the investigator.
- ATM-AVI + Metronidazole: High AVI Dose Cohort: Participants received ATM-AVI IV infusion in following manner (1. normal renal function or mild renal impairment [CrCl >50mL/min] : 500 mg ATM plus 167 mg AVI over 30 minutes as loading dose, followed by maintenance infusions of 1500 mg ATM plus 500 mg AVI, over a 3 hour period every 6 hours; 2. moderate renal impairment [CrCl 31-50 ml/min]: 500 mg ATM plus 167 mg AVI over 30 minutes as loading dose, followed by IV extended loading infusion of 1500 mg ATM plus 500 mg AVI over 3 hour, followed by maintenance infusions of 750 mg ATM plus 250 mg AVI, over 3 hour period every 6 hours) along with 1 hour IV infusion of 500 mg metronidazole, every 8 hrs after first ATM-AVI maintenance infusion. All treatments were administered for minimum 5 days and up to maximum of 14 days. All study therapies could be discontinued (after at least 5 full days of IV therapy) at the discretion of the investigator.
Period: Overall Study
Arm/Group | Aztreonam-Avibactam(ATM-AVI)+Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Started | 17 | 23
Treated | 16 | 18
Completed | 12 | 16
Not Completed | 5 | 7
Not completed — Enrolled but not treated | 1 | 5
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (MITT) population included all enrolled participants who received any amount of study drug.
Groups:
- ATM-AVI+ Metronidazole:Low AVI Dose Cohort: Participants with normal renal function or mild renal impairment (CrCl > 50 mL/min), received IV infusion of 500 mg ATM plus 137 mg AVI over 30 minutes as loading dose, followed by maintenance infusions of 1500 mg ATM plus 410 mg AVI, over a 3 hour period every 6 hours, for a minimum of 5 days and up to maximum of 14 days. Participants also received 1 hour IV infusion of 500 mg metronidazole, every 8 hrs after first ATM-AVI maintenance infusion for a minimum of 5 days and up to maximum of 14 days. All study therapies could be discontinued (after at least 5 full days of IV therapy) at the discretion of the investigator.
- Total: Total of all reporting groups
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.00 (12.47) | 53.06 (14.25) | 51.15 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 12 | 14 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 17 | 30
  Other | 1 | 0 | 1
  Unknown | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Sparse Sampling at Day 1, 0 hr
Description: All participants were to have sparse pharmacokinetics (PK) sampling on Day 1; the first sequentially enrolled 25 participants in study were to have intensive PK sampling on Day 4 while the remaining participants were to have sparse sampling on Day 4. Data was summarized only for observations above lower limit of quantification (LLOQ). LLOQ for ATM was 0.1 microgram per milliliter (mcg/ml).
Time Frame: Predose (0 hr) on Day 1
Population: PK population included all participants who had at least 1 plasma concentration data assessment available for ATM-AVI. Here, Overall number of participants analyzed signifies participants who had observations above LLOQ.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 1 | 0
microgram per milliliter (mcg/mL) | 0.1 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |

2. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Sparse Sampling at Day 1, 0.42 hr
Description: All participants were to have sparse PK sampling on Day 1; the first sequentially enrolled 25 participants in study were to have intensive PK sampling on Day 4 while the remaining participants were to have sparse sampling on Day 4. Data was summarized only for observations above LLOQ. LLOQ for ATM was 0.1 mcg/ml.
Time Frame: 0.42 hr Post dose on Day 1
Population: The PK population included all participants who had at least 1 plasma concentration data assessment available for ATM-AVI.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
mcg/mL | 39.0 (262.0) | 39.4 (58.1)

3. Primary Outcome: Plasma Concentrations of Aztreonam (ATM): Sparse Sampling at Day 1, 3.25 hr
Description: as for outcome 2
Time Frame: 3.25 hr Post dose on Day 1
Population: The PK population included all participants who had at least 1 plasma concentration data assessment available for ATM-AVI. Here, Overall number of participants analyzed signifies participants who had observations above LLOQ.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
mcg/mL | 55.7 (16.0) | 58.5 (36.3)

4. Primary Outcome: Plasma Concentrations of Aztreonam (ATM): Sparse Sampling at Day 1, 5 hr
Description: as for outcome 2
Time Frame: 5 hr Post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- ATM-AVI + Metronidazole: Low AVI Dose Cohort: Participants with normal renal function or mild renal impairment (CrCl > 50 mL/min), received IV infusion of 500 mg ATM plus 137 mg AVI over 30 minutes as loading dose, followed by maintenance infusions of 1500 mg ATM plus 410 mg AVI, over a 3 hour period every 6 hours, for a minimum of 5 days and up to maximum of 14 days. Participants also received 1 hour IV infusion of 500 mg metronidazole, every 8 hrs after first ATM-AVI maintenance infusion for a minimum of 5 days and up to maximum of 14 days. All study therapies could be discontinued (after at least 5 full days of IV therapy) at the discretion of the investigator.
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
mcg/mL | 28.8 (23.9) | 31.5 (50.8)

5. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 1, 0 hr
Description: All participants were to have sparse PK sampling on Day 1; the first sequentially enrolled 25 participants in study were to have intensive PK sampling on Day 4 while the remaining participants were to have sparse sampling on Day 4. Data was summarized only for observations above LLOQ. LLOQ for AVI was 10 nanogram per milliliter (ng/ml).
Time Frame: Predose (0 hr) on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 1 | 0
nanogram per milliliter (ng/mL) | 24.9 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |

6. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 1, 0.42 hr
Description: All participants were to have sparse PK sampling on Day 1; the first sequentially enrolled 25 participants in study were to have intensive PK sampling on Day 4 while the remaining participants were to have sparse sampling on Day 4. Data was summarized only for observations above LLOQ. LLOQ for AVI was 10 ng/ml.
Time Frame: 0.42 hr Post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
ng/mL | 7852.6 (279.2) | 9801.5 (61.8)

7. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 1, 3.25 hr
Description: as for outcome 6
Time Frame: 3.25 hr Post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
ng/mL | 9976.5 (25.8) | 12982.7 (49.7)

8. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 1, 5 hr
Description: as for outcome 6
Time Frame: 5 hr Post dose on Day 1
Population: PK population: all participants who had at least 1 plasma concentration data available for ATM-AVI. Here, Overall number of participants analyzed signifies participants who had observations above LLOQ. Intensive rather than sparse sampling was conducted for all participants in low AVI dose cohort(Cohort 1)on Day4 and hence sparse data not reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 17
ng/mL | 4086.6 (35.3) | 5549.0 (76.6)

9. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Sparse Sampling at Day 4, 0 hr
Description: as for outcome 2
Time Frame: Predose (0 hr) on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
mcg/mL | 19.7 (29.0)

10. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Sparse Sampling at Day 4, 2.75 hr
Description: as for outcome 2
Time Frame: 2.75 hr Post dose on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
mcg/mL | 46.4 (19.5)

11. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Sparse Sampling at Day 4, 5 hr
Description: as for outcome 2
Time Frame: 5 hr Post dose on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
mcg/mL | 16.5 (37.3)

12. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 4, 0 hr
Description: as for outcome 6
Time Frame: Predose (0 hr) on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
ng/mL | 4048.8 (24.3)

13. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 4, 2.75 hr
Description: as for outcome 6
Time Frame: 2.75 hr Post dose on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
ng/mL | 9073.6 (24.2)

14. Primary Outcome: Plasma Concentration of Avibactam (AVI): Sparse Sampling at Day 4, 5 hr
Description: as for outcome 6
Time Frame: 5 hr Post dose on Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 8
ng/mL | 2745.7 (40.5)

15. Primary Outcome: Plasma Concentration Aztreonam (ATM): Intensive Sampling at Day 4, 0 hr
Description: as for outcome 2
Time Frame: Predose (0 hr) on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 18.3 (71.2) | 20.3 (88.5)

16. Primary Outcome: Plasma Concentration Aztreonam (ATM): Intensive Sampling at Day 4, 0.5 hr
Description: as for outcome 2
Time Frame: 0.5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Higher AVI Dose (Cohorts 2+3): Participants with cIAI, having CrCl >50mL/min, received ATM plus AVI at loading dose of 500mg ATM plus higher dose AVI(167mg), IV for 30minute period, followed by maintenance infusions of 1500mg ATM plus 500mg AVI, over 3hr period every 6hrs, for maximum of 14days. Participants with CrCl 31-50mL/min, either received loading dose consistent with Cohort 1, followed by extended loading infusion of 1500mg ATM plus 410mg AVI over 3hr period, followed by(3hrs after stop of second loading infusion) maintenance infusion of 750mg ATM plus 205mg AVI over 3hr period(administered every 6hrs) or loading dose consistent with higher AVI dose in Cohort 2, followed by extended loading infusion of 1500mg ATM plus 500mg AVI over 3hrperiod, followed by maintenance infusion of 750mg ATM plus 250mg AVI over 3hr period(administered every 6hrs). Participants also received 500mg metronidazole infused over 1hr every 8hrs after first ATM-AVI maintenance infusion(Day5 to Day14) at investigator's discretion.
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | Higher AVI Dose (Cohorts 2+3)
Number analyzed (Participants) | 12 | 8
mcg/mL | 37.6 (194.0) | 33.8 (46.0)

17. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 1 hr
Description: as for outcome 2
Time Frame: 1 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 41.2 (53.5) | 43.0 (44.7)

18. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 2 hr
Description: as for outcome 2
Time Frame: 2 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 49.6 (42.5) | 53.6 (44.7)

19. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 3 hr
Description: as for outcome 2
Time Frame: 3 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 53.6 (72.0) | 54.7 (42.1)

20. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 3.25 hr
Description: as for outcome 2
Time Frame: 3.25 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
mcg/mL | 45.8 (36.7) | 47.3 (49.8)

21. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 3.5 hr
Description: as for outcome 2
Time Frame: 3.5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
mcg/mL | 42.9 (37.9) | 43.2 (52.1)

22. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 3.75 hr
Description: as for outcome 2
Time Frame: 3.75 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
mcg/mL | 39.5 (41.8) | 38.5 (57.6)

23. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 4 hr
Description: as for outcome 2
Time Frame: 4 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
mcg/mL | 34.2 (44.2) | 36.6 (63.3)

24. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 5 hr
Description: as for outcome 2
Time Frame: 5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 23.8 (56.1) | 26.4 (76.8)

25. Primary Outcome: Plasma Concentration of Aztreonam (ATM): Intensive Sampling at Day 4, 6 hr
Description: as for outcome 2
Time Frame: 6 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | Higher AVI Dose (Cohorts 2+3)
Number analyzed (Participants) | 13 | 8
mcg/mL | 22.2 (149.8) | 19.0 (97.1)

26. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 0 hr
Description: as for outcome 6
Time Frame: Predose (0 hr) on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 2516.2 (85.6) | 3184.3 (137.5)

27. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 0.5 hr
Description: as for outcome 6
Time Frame: 0.5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
ng/mL | 6374.4 (215.4) | 7140.3 (69.3)

28. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 1 hr
Description: as for outcome 6
Time Frame: 1 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 7369.8 (59.2) | 9435.7 (64.4)

29. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 2 hr
Description: as for outcome 6
Time Frame: 2 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 8885.4 (48.5) | 11668.0 (59.5)

30. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 3 hr
Description: as for outcome 6
Time Frame: 3 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 9820.4 (100.1) | 11903.2 (62.6)

31. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 3.25 hr
Description: as for outcome 6
Time Frame: 3.25 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
ng/mL | 8009.9 (38.7) | 9631.5 (66.0)

32. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 3.5 hr
Description: as for outcome 6
Time Frame: 3.5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
ng/mL | 7095.8 (43.9) | 8545.4 (83.8)

33. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 3.75 hr
Description: as for outcome 6
Time Frame: 3.75 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
ng/mL | 6340.3 (50.3) | 7227.1 (88.4)

34. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 4 hr
Description: as for outcome 6
Time Frame: 4 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 8
ng/mL | 5258.7 (49.9) | 6727.6 (94.2)

35. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 5 hr
Description: as for outcome 6
Time Frame: 5 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 3300.0 (59.7) | 4300.3 (120.9)

36. Primary Outcome: Plasma Concentration of Avibactam (AVI): Intensive Sampling at Day 4, 6 hr
Description: as for outcome 6
Time Frame: 6 hr Post dose on Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 3275.7 (205.4) | 2879.2 (140.1)

37. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Aztreonam (ATM): Intensive Sampling at Day 4
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: The PK population included all participants who had at least 1 plasma concentration data assessment available for ATM-AVI. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
mcg/mL | 62.5 (146.9) | 55.4 (42.6)

38. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avibactam (AVI): Intensive Sampling at Day 4
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
ng/mL | 11552.4 (164.5) | 12116.2 (61.2)

39. Primary Outcome: Time of Observed Maximum Concentration (Tmax) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Median (Full Range); unit: hours
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hours
  ATM | 2.9 [0.5 to 3.5] | 2.4 [2.0 to 3.0]
  AVI | 2.9 [0.5 to 3.8] | 2.8 [2.0 to 3.3]

40. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours (AUC[0-6]) for Aztreonam (ATM): Intensive Sampling at Day 4
Description: AUC(0-6) was defined as the area under the plasma concentration-time curve from time zero up to the six hours postdose.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (hr*mcg/mL)
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hour*microgram/milliliter (hr*mcg/mL) | 235.2 (60.6) | 234.7 (54.6)

41. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours (AUC[0-6]) for Avibactam (AVI): Intensive Sampling at Day 4
Description: AUC(0-6) was defined as the area under the plasma concentration-time curve from time zero up to the six hours postdose.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hour*nanogram per milliliter (hr*ng/mL) | 40437.0 (74.0) | 47477.5 (79.2)

42. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to the Last Measured Concentration (AUC[0-last]) for Aztreonam (ATM): Intensive Sampling at Day 4
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve from time zero up to the time of the last measurable concentration.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hr*mcg/mL | 235.9 (60.4) | 234.3 (54.7)

43. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to the Last Measured Concentration (AUC[0-last]) for Avibactam (AVI): Intensive Sampling at Day 4
Description: as for outcome 42
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hr*ng/mL | 40539.5 (73.8) | 47422.2 (79.3)

44. Primary Outcome: Time of Last Measured Concentration (Tlast) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Median (Full Range); unit: hours
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
hours
  ATM | 6.0 [6.0 to 6.5] | 6.0 [5.9 to 6.0]
  AVI | 6.0 [6.0 to 6.5] | 6.0 [5.9 to 6.0]

45. Primary Outcome: Plasma Elimination Half-life (t1/2) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Description: Plasma elimination half-life was defined as time measured for the plasma concentration of ATM and AVI to decrease by one half of its initial concentration.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 11 | 8
hours
  ATM | 2.3 (1.06) | 2.8 (2.05)
  AVI | 1.8 (0.59) | 2.2 (1.85)

46. Primary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Description: Apparent volume of distribution at steady state was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 11 | 8
liter
  ATM | 20.3 (16.9) | 19.6 (31.8)
  AVI | 26.0 (22.0) | 23.7 (29.7)

47. Primary Outcome: Volume of Distribution (Vz) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Standard Deviation); unit: liter
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 11 | 8
liter
  ATM | 21.4 (15.3) | 21.6 (24.1)
  AVI | 28.2 (20.4) | 27.4 (20.6)

48. Primary Outcome: Apparent Clearance (CL) of Aztreonam (ATM) and Avibactam (AVI): Intensive Sampling at Day 4
Description: Clearance of a drug was measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 8
liter/hour
  ATM | 6.4 (35.4) | 6.4 (35.5)
  AVI | 10.1 (42.6) | 10.5 (41.4)

49. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAEs was an AE resulting in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; or was an important medical event which may jeopardise the participants or require medical intervention to prevent one of the above outcomes. Treatment-emergent were events between first infusion of study drug and up to late follow-up (LFU) visit (20 to 24 days after last infusion). AEs included both non-serious AEs and SAEs.
Time Frame: From first dose of study drug up to the LFU visit (up to maximum of 38 days)
Population: The safety analysis included all enrolled participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
Participants
  AEs | 11 | 12
  SAEs | 4 | 5

50. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: QT value: greater than or equal to (>=) 450 milliseconds (msec), >=480 msec, >=500 msec, >=500 and increase from baseline >=60 msec. Increase from baseline in QT: >=30 msec, >=60 msec. Decrease from baseline in QT: >=30 msec, >=60 msec. QTcB value: >=450 msec, >=480 msec, >=500 msec, >=500 and increase from baseline >=60 msec. Increase from baseline in QT interval using Bazett's correction (QTcB) value: >=30 msec, >=60 msec. Decrease from baseline in QTcB: >=30 msec, >=60 msec. QT interval using Fridericia's correction (QTcF) value: >=450 msec, >=480 msec, >=500 msec, >=500 and increase from baseline >=60 msec. Increase from baseline in QTcF value: >=30 msec, >=60 msec. Decrease from baseline in QTcF value: >=30 msec, >=60 msec. EOT (end of treatment) visit occurred within 24 hours after last infusion.
Time Frame: Baseline up to EOT (up to a maximum of 15 days)
Population: The safety analysis included all enrolled participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
Participants
  QT value >=450 | 2 | 0
  QT value >=480 | 2 | 0
  QT value >=500 | 2 | 0
  QT value >=500 and increase from baseline >=60 | 1 | 0
  Increase in QT >=30 | 6 | 4
  Increase in QT>=60 | 2 | 1
  Decrease in QT >=30 | 1 | 1
  Decrease in QT>=60 | 0 | 1
  QTcB value >=450 | 5 | 1
  QTcB value >=480 | 2 | 0
  QTcB value >=500 | 1 | 0
  QTcB value >=500 and increase from baseline >=60 | 0 | 0
  Increase in QTcB >=30 | 3 | 1
  Increase in QTcB >=60 | 0 | 1
  Decrease in QTcB >=30 | 2 | 1
  Decrease in QTcB >=60 | 0 | 0
  QTcF value >=450 | 4 | 0
  QTcF value >=480 | 2 | 0
  QTcF value >=500 | 1 | 0
  QTcF value >=500 and increase from baseline >=60 | 0 | 0
  Increase in QTcF >=30 | 3 | 2
  Increase in QTcF >=60 | 0 | 0
  Decrease in QTcF >=30 | 0 | 1
  Decrease in QTcF >=60 | 0 | 0

51. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities in Hematology Parameters
Description: Criteria for abnormality: Hemoglobin, hematocrit, erythrocytes less than(<) 0.7*lower limit of normal [LLN] and (&) greater than (>) 30 percent (%) below baseline [BB]; >1.3*upper limit of normal [ULN] & >30% above baseline [AB], leukocytes <0.65*LLN & >60% BB; >1.6* ULN & >100% AB; platelets <0.65*LLN & >50% BB; >1.5*ULN & >100% AB; neutrophils <0.65*LLN & >75% BB; >1.6*ULN & >100% AB, lymphocytes <0.25*LLN & >75%BB; >1.5*ULN & >100% AB, basophils, eosinophils, monocytes>4.0*ULN & >300% AB. LFU visit occurred within 20 to 24 days after last infusion.
Time Frame: Baseline up to LFU visit (up to maximum of 38 days)
Population: The safety analysis included all enrolled participants who received any amount of study drug. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 17
Participants
  Hemoglobin: <0.7*LLN&>30% BB | 0 | 0
  Hemoglobin: >1.3*ULN&>30% AB | 0 | 0
  Hematocrit: <0.7*LLN&>30% BB | 0 | 0
  Hematocrit:>1.3*ULN&>30% AB | 0 | 0
  Erythrocytes:<0.7*LLN&>30% BB | 0 | 0
  Erythrocytes: >1.3*ULN&>30% AB | 0 | 0
  Leukocytes: <0.65*LLN&>60%BB | 0 | 0
  Leukocytes:>1.6* ULN&>100%AB | 1 | 0
  Platelets: <0.65*LLN&>50%BB | 0 | 0
  Platelets: >1.5*ULN&>100% AB | 1 | 5
  Neutrophils:<0.65*LLN&>75% BB | 0 | 0
  Neutrophils: >1.6*ULN & >100% AB | 1 | 1
  Lymphocytes: <0.25*LLN&>75%BB | 0 | 0
  Lymphocytes: >1.5*ULN&>100%AB | 0 | 0
  Basophils: >4.0*ULN&>300% AB | 0 | 0
  Eosinophils: >4.0*ULN&>300% AB | 0 | 0
  Monocytes: >4.0*ULN&>300% AB | 0 | 0

52. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities in Clinical Chemistry Paramteres
Description: Criteria for abnormality: aspartate aminotransferase, alanine aminotransferase >3.0*ULN & >100% AB, alkaline phosphatase <0.5 *LLN & >80% BB&; >3.0*ULN & >100% AB; bilirubin >1.5*ULN & >100% AB; direct bilirubin >2.0*ULN & >150% AB; protein <0.5*LLN & >50%BB; >1.5*ULN & >50% AB, albumin <0.5*LLN & >50% BB; >1.5*ULN & >50% AB, urea nitrogen <0.2* LLN & >100% BB; >3.0*ULN & >200% AB, creatinine >2.0*ULN & >100% AB, sodium <0.85*LLN & >10% BB;>1.1*ULN &>10% AB; potassium <0.8*LLN &>20% BB; >1.2*ULN &>20% AB, chloride <0.8*LLN &>20% BB;>1.2*ULN & >20% AB, calcium <0.7*LLN & >30% BB; >1.3*ULN & >30% AB, phosphate <0.5*LLN & >50% BB; >3.0*ULN & >200% AB, bicarbonate <0.7*LLN & >40% BB; >1.3*ULN & >40% AB, glucose <0.6*LLN & >40% BB, >3.0*ULN & >200% AB. LFU visit occurred within 20 to 24 days after last infusion.
Time Frame: Baseline up to LFU visit (up to maximum of 38 days)
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 13 | 17
Participants
  Aspartate aminotransferase: >3.0*ULN&>100% AB | 1 | 0
  Alanine aminotransferase:>3.0x ULN | 2 | 2
  Alkaline phosphatase: <0.5 *LLN&>80% BB& | 0 | 0
  Alkaline phosphatase:>3.0*ULN&>100%AB | 0 | 0
  Bilirubin: >1.5*ULN&>100%AB | 0 | 0
  Direct Bilirubin : >2.0*ULN&>150% AB | 0 | 0
  Protein: <0.5*LLN &>50%BB | 0 | 0
  Protein: >1.5*ULN&>50% AB | 0 | 0
  Albumin: <0.5*LLN&>50%BB | 0 | 0
  Albumin: >1.5*ULN&>50%AB | 0 | 0
  Urea nitrogen: <0.2* LLN&>100%BB | 0 | 0
  Urea nitrogen: >3.0*ULN&>200%AB | 0 | 0
  Creatinine: >2.0*ULN&>100%AB | 0 | 0
  Sodium: < 0.85*LLN&>10%BB | 0 | 0
  Sodium: >1.1*ULN&>10%AB | 0 | 0
  Potassium: <0.8*LLN&>20%BB | 1 | 1
  Potassium: >1.2*ULN&>20%AB | 0 | 0
  Chloride: <0.8*LLN&>20%BB | 0 | 0
  Chloride: >1.2*ULN&>20%AB | 0 | 0
  Calcium: <0.7*LLN&>30% BB | 0 | 0
  Calcium: >1.3*ULN&>30%AB | 0 | 0
  Phosphate: <0.5*LLN&>50% BB | 0 | 0
  Phosphate: >3.0*ULN&>200% AB | 0 | 0
  Bicarbonate: <0.7*LLN&>40% BB | 0 | 0
  Bicarbonate: >1.3*ULN&>40%AB | 0 | 0
  Glucose: <0.6*LLN&>40% BB | 0 | 0
  Glucose: >3.0*ULN&>200%AB | 0 | 0

53. Primary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital sign parameters included: Supine systolic blood pressure (millimeters of mercury [mmHg]), Supine diastolic blood pressure (mmHg), Heart rate (beats per minute), Respiratory rate (breaths per minute) and body temperature (degree celsius). Criteria for clinical significance in vital signs was based on investigator's assessment. LFU visit occurred within 20 to 24 days after last infusion.
Time Frame: From first dose of study drug up to LFU visit (up to maximum of 38 days)
Population: The safety analysis included all enrolled participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
Participants
  Supine systolic blood pressure | 0 | 0
  Supine diastolic blood pressure | 0 | 0
  Heart rate | 0 | 0
  Respiratory rate | 0 | 1
  Temperature | 0 | 0

54. Primary Outcome: Number of Participants With Clinical Significant Physical Examination Findings : MITT Population
Description: Physical examinations included an assessment of abdomen, cardiovascular, general appearance, head, eyes, ears, nose, lymph nodes, skin, musculoskeletal, neurological, respiratory systems and other (edemas). Clinically significant abnormality in physical examination was based on investigator's assessment. LFU visit occured within 20 to 24 days after last infusion.
Time Frame: From first dose of study drug up to the LFU visit (up to maximum of 38 days)
Population: The MITT population included all enrolled participants who received any amount of study drug. Here, 'number analysed' = Participants evaluable for this outcome measure at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
Participants
  Abdomen: number analyzed (Participants) | 13 | 17
  Abdomen | 1 | 0
  Cardiovascular: number analyzed (Participants) | 13 | 17
  Cardiovascular | 0 | 0
  General appearance: number analyzed (Participants) | 13 | 17
  General appearance | 0 | 1
  Head, Eyes, Ears, Nose: number analyzed (Participants) | 13 | 17
  Head, Eyes, Ears, Nose | 0 | 0
  Lymph nodes: number analyzed (Participants) | 13 | 17
  Lymph nodes | 0 | 0
  Musculoskeletal system: number analyzed (Participants) | 13 | 17
  Musculoskeletal system | 0 | 0
  Neurological system: number analyzed (Participants) | 13 | 17
  Neurological system | 0 | 0
  Other: number analyzed (Participants) | 3 | 2
  Other | 0 | 1
  Respiratory system: number analyzed (Participants) | 13 | 17
  Respiratory system | 0 | 1
  Skin: number analyzed (Participants) | 13 | 17
  Skin | 0 | 0

55. Secondary Outcome: Percentage of Participants With Clinical Cure at Test of Cure (TOC) Visit: MITT Population
Description: Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of the index infection (cIAI) such as no further antimicrobial therapy, drainage, or surgical intervention is necessary and does not meet any of the failure criteria. Failure: death related to intra-abdominal infection; received treatment with additional antibiotics for ongoing symptoms of cIAI; previously met criteria for failure; persisting or recurrent infection within the abdomen; post-surgical wound infections included an open wound with signs of local infection such as purulent exudates, erythema, or warmth that requires additional antibiotics and/or non-routine wound care. TOC visit occurred up to a maximum of 28 days after first dose.
Time Frame: Test of Cure Visit (up to a maximum of 28 days)
Population: The MITT population included all enrolled participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
percentage of participants | 62.5 [35.4 to 84.8] | 55.6 [30.8 to 78.5]

56. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit: Microbiologically Modified Intent-to-Treat (mMITT) Population
Description: as for outcome 55
Time Frame: Test of Cure Visit (up to a maximum of 28 days)
Population: The mMITT population included all enrolled participants who had any amount of study drug and had a diagnosis of cIAI (that is,met inclusion criterion ) and an intraabdominal pathogen at baseline. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATM-AVI + Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 11
percentage of participants | 66.7 [34.9 to 90.1] | 54.5 [23.4 to 83.3]

57. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours [AUC(0-6)] of Aztreonam (ATM) for Participants With Clinical Cure and Failure at TOC Visit: Intensive Sampling at Day 4 (MITT Population)
Description: AUC(0-6): area under the plasma concentration-time curve from time 0 upto the 6hrs. Clinical cure;complete resolution or significant improvement of signs and symptoms of the index infection(cIAI)such as no further antimicrobial therapy, drainage, or surgical intervention necessary and does not meet any of failure criteria. Failure: death related to intra-abdominal infection; received treatment with additional antibiotics for ongoing symptoms of cIAI; previously met criteria for failure; persisting or recurrent infection within abdomen; post-surgical wound infections included an open wound with signs of local infection such as purulent exudates, erythema, or warmth that requires additional antibiotics and/or non-routine wound care. Data of AUC(0-6) based on intensive sampling at Day4, is reported in this outcome separately and only for those participants who had clinical response of cure and failure at TOC Visit. TOC visit occurred up to a maximum of 28 days after first dose.
Time Frame: Plasma samples collection for AUC0-6 at: predose, 0.5 1, 2, 3, 3.25, 3.5, 3.75, 4, 5 and 6 hour postdose on Day 4 assessed for participants with cure and failure at Test of Cure Visit (up to a maximum of 28 days)
Population: The MITT population included all enrolled participants who received any amount of study drug. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified categories. AUC0-6 was assessed on Day 4 and presented in this OM, only for those participants who had clinical cure or failure at TOC visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
hr*mcg/mL
  Clinical Cure: number analyzed (Participants) | 10 | 4
  Clinical Cure | 226.0 (43.0) | 218.7 (28.5)
  Clinical Failure: number analyzed (Participants) | 3 | 2
  Clinical Failure | 268.9 (88.3) | 169.8 (14.9)

58. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours [AUC(0-6)] of Avibactam (AVI) for Participants With Clinical Cure and Failure at TOC Visit: Intensive Sampling at Day 4 (MITT Population)
Description: as for outcome 57
Time Frame: as for outcome 57
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 16 | 18
hr*ng/mL
  Clinical Cure: number analyzed (Participants) | 10 | 4
  Clinical Cure | 38003.8 (45.7) | 40314.0 (36.1)
  Clinical Failure: number analyzed (Participants) | 3 | 2
  Clinical Failure | 49730.0 (100.1) | 34633.7 (10.2)

59. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours [AUC(0-6)] of Aztreonam (ATM) for Participants With Clinical Cure and Failure at TOC Visit: Intensive Sampling at Day 4 (mMITT Population)
Description: as for outcome 57
Time Frame: as for outcome 57
Population: mMITTpopulation set was used in this analysis. Here, 'Number analyzed' = participants evaluable for this outcome measure at specified categories. AUC0-6 was assessed on Day 4 and presented in this OM, only for those participants who had clinical cure or failure at TOC visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | ATM-AVI+ Metronidazole:Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 11
hr*mcg/mL
  Clinical Cure: number analyzed (Participants) | 8 | 1
  Clinical Cure | 245.3 (41.4) | 292.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Clinical Failure: number analyzed (Participants) | 2 | 0
  Clinical Failure | 378.0 (77.0) |

60. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero up to 6 Hours [AUC(0-6)] of Avibactam (AVI) for Participants With Clinical Cure and Failure at TOC Visit: Intensive Sampling at Day 4 (mMITT Population)
Description: as for outcome 57
Time Frame: as for outcome 57
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- ATM-AVI+ Metronidazole: Low AVI Dose Cohort: Participants with normal renal function or mild renal impairment (CrCl > 50 mL/min), received IV infusion of 500 mg ATM plus 137 mg AVI over 30 minutes as loading dose, followed by maintenance infusions of 1500 mg ATM plus 410 mg AVI, over a 3 hour period every 6 hours, for a minimum of 5 days and up to maximum of 14 days. Participants also received 1 hour IV infusion of 500 mg metronidazole, every 8 hrs after first ATM-AVI maintenance infusion for a minimum of 5 days and up to maximum of 14 days. All study therapies could be discontinued (after at least 5 full days of IV therapy) at the discretion of the investigator.
Arm/Group | ATM-AVI+ Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
Number analyzed (Participants) | 12 | 11
hr*ng/mL
  Clinical Cure: number analyzed (Participants) | 8 | 1
  Clinical Cure | 42401.9 (41.9) | 60302.1 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Clinical Failure: number analyzed (Participants) | 2 | 0
  Clinical Failure | 75509.9 (84.3) |

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to the LFU visit (up to maximum of 38 days)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Analysis was performed on safety population.
Arm/Group | ATM-AVI+ Metronidazole: Low AVI Dose Cohort | ATM-AVI + Metronidazole: High AVI Dose Cohort
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/18
Serious Adverse Events (participants affected / at risk) | 4/16 | 5/18
Other Adverse Events (participants affected / at risk) | 10/16 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATM-AVI+ Metronidazole: Low AVI Dose Cohort (N=16) | ATM-AVI + Metronidazole: High AVI Dose Cohort (N=18)
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATM-AVI+ Metronidazole: Low AVI Dose Cohort (N=16) | ATM-AVI + Metronidazole: High AVI Dose Cohort (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Chronic hepatitis C (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 7 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results

DOCUMENTS (2):
  • Study Protocol (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02655419/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT02655419/SAP_001.pdf